CLINICAL TRIAL: NCT01825577
Title: Exploring the Use of Transdermal Methylphenidate to Reduce Fall Risk in Patients With Dementia.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Administrative Reasons
Sponsor: St. Louis University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23014
Record Dates: First submitted 2013-03-13; First posted 2013-04-05 (Estimated); Results first posted 2016-08-19 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2016-08

CONDITIONS: Dementia; Accidental Falls; Apathy
Keywords: Alzheimer Dementia; Gait
MeSH Terms: conditions — Dementia; Lethargy; Alzheimer Disease | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transdermal Methylphenidate (Experimental): 2 Weeks of once daily 10mg Transdermal Methylphenidate followed by 2 weeks of once daily 15mg Transdermal Methylphenidate. Patch will be worn for approximately 7-10hrs each day.
  Interventions: Drug: Transdermal Methylphenidate

INTERVENTIONS:
Drug: Transdermal Methylphenidate — 2 Weeks of once daily 10mg Transdermal Methylphenidate followed by 2 weeks of once daily 15mg Transdermal Methylphenidate. Patch will be worn for approximately 7-10hrs each day.
  Other Names: Daytrana

SUMMARY:
Falls in the elderly are a very common and serious health problem with devastating consequences. Those with dementia are 5 times more likely to experience falls than older people without significant cognitive impairment. Despite a growing awareness and the use of available treatments, the number of falls and fall related injuries continue to increase. It is important to develop more effective treatments to help reduce the number of falls and prevent injury. The assessments used in this study determine fall risk which predicts the likelihood of falls in the future.

This study will evaluate the possible role of Methylphenidate, Ritalin, in preventing falls and improving symptoms of apathy, or indifference. Methylphenidate is FDA approved for the treatment of ADHD but is not currently approved by the FDA for preventing falls or improving apathy(lack of interest) in the elderly. The methylphenidate used in this study will be absorbed through the skin by wearing a small patch near the hip area.

The specific primary aim of this open label study is to determine if use of transdermal Methylphenidate (t-MPH) causes a reduction in fall risk in patients with dementia.

The hypotheses to be tested is that after receiving t-MPH for 4 weeks, subjects will show improvement in gait and mobility assessment scores when compared to gait and mobility scores at screening.

DETAILED DESCRIPTION:
This is an open label pilot study; consenting subjects with dementia and identified as a fall risk, who meet inclusion criteria will undergo 3 phases of involvement. Phase 1 is a 1 week period before initiating study drug. Phase 2 is a 2 week treatment period with 10mg of Transdermal Methylphenidate. Phase 3 is the final two week treatment period with 15mg of Transdermal Methylphenidate.

Measurements obtained at each phase will include:

Vital Signs (blood pressure and pulse rate) weight , Timed Get Up and Go Test (TUG) , Tinetti Performance Oriented Mobility Assessment (POMA), Clinical Apathy Evaluation Scale (AES-C) and the St. Louis University Mental Status Examination (SLUMS).

The primary endpoint is the change in TUG and POMA scores at end of phase 3 compared to beginning of phase 2

Falls are a cause of substantial morbidity and mortality in patients with dementia and occur at twice the rate of older adults without cognitive impairment. The consequences of falls in older adults with dementia are serious; fallers with cognitive problems are approximately five times as likely to be admitted to institutional care as people with cognitive problems who do not fall.[3] They are also at high risk of major fall-related injuries such as fractures and head injuries that increase mortality risk.

Walking requires paying attention to various environmental features and recovering from postural variations to avoid stumbles or falls. Consequently, deficits in attention and executive function are independently associated with risk of postural instability, impairment in activities of daily living, and fall risk.

Executive function refers to higher cognitive processes that allocate attention among tasks and a critical cognitive resource for normal walking. Lower scores on executive function measures are associated with both dementia and a higher fall risk. Although significant progress towards understanding the factors involved in falls has been made, the number of falls and fall related injuries continue to increase.

Changes in aging demographics are expected to dramatically increase the aging population and dementia prevalence, underscoring the importance of developing more effective fall prevention strategies.

Recent studies have shown that improving certain aspects of cognition, specifically attention and executive function, in older adults can improve mobility decline and risk of falls. Particularly in cognitively impaired individuals, this may be critical to reducing fall risk.

Why Methylphenidate?

Pharmacological properties of psychostimulants, such as methylphenidate (MPH), are known to increase executive function. Methylphenidate was chosen because of the studies demonstrating the safe use of MPH for treatment of depression and apathy in the cognitively impaired elderly and the well-studied effects of MPH on executive function and attention in children and adults with ADHD.

Also a small study published in April 2008 in J Am Geriatric Society, evaluated the use of methylphenidate in reducing fall risk among community living older adults. The study concluded that among study subjects receiving methylphenidate, significant improvement in mobility and gait assessments were observed as well as drug tolerability.

The basis for our study is to further explore the pharmacotherapeutic role of Transdermal-MPH in reducing fall risk in dementia patients.

Mobility and gait assessment performance is strongly correlated with fall risk. Therefore we will use subject's scores before, during and after medication administration to measure response and evaluate use as a fall prevention strategy.

ELIGIBILITY:
Inclusion Criteria:

1. 65- 95 years of age
2. Ability to ambulate (may use walking aid)
3. Male or Female
4. Clinical diagnosis of Dementia
5. Identified as fall risk by nursing staff

Exclusion Criteria:

1. Clinically significant musculoskeletal, cardiovascular or respiratory diseases.
2. Clinically significant vestibular disorder
3. History of significant head trauma
4. Any medically unstable condition, as determined by the PI that would expose patient to potential harm.
5. Patients taking medications that may interact with MPH, as determined by manufacture's package insert.

   Including but not limited to: Warfarin, anticonvulsants, MAOIs, alpha2-agonists, tri-cyclic antidepressants.
6. Legally Blind
7. History of seizures,
8. Poorly controlled hypertension, cardiac arrhythmia or cardiovascular disease, heart failure.
9. Known or suspected allergy to MPH or similar compounds
10. Glaucoma
11. Motor tics
12. History of significant agitation or anxiety
13. Family history of Tourette's syndrome
14. History of significant anxiety
15. History of significant agitation
16. History of significant tension.

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George T Grossberg, M.D., Principal Investigator — Saint Louis University School of Medicine Department of Neurology and Psychiatry; Ahmed A Baig, M.D., Principal Investigator — Saint Louis University School of Medicine Department of Neurology and Psychiatry
Locations (1):
- Delmar Gardens, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Transdermal Methylphenidate: 1. Age 65 yrs and above
  2. Ability to ambulate (may use walking aid)
  3. Male or Female
  4. Clinical diagnosis of probable Alzheimer's Disease
  5. AES score >40
  6. Identified as fall risk by nursing staff
Period: Overall Study
Arm/Group | Single Arm Transdermal Methylphenidate
Started | 14
Completed | 6
Not Completed | 8
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 1
Not completed — Withdrawn by family members | 2
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: 1. Age 65yrs and above
  2. Ability to ambulate (may use walking aid)
  3. Male or Female
  4. Clinical diagnosis of probable Alzheimer's Disease
  5. AES score >40
  6. Identified as fall risk by nursing staff
Arm/Group | Single Arm
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Timed Get Up and Go Test - Measure of Mobility
Description: Timed Get Up and Go Test (TUG), is used to evaluate the ability to walk by measuring the time it takes to rise from a chair, walk 10 feet, turn around, walk back to the chair, and sit down. The TUG test takes less than 5 minutes to complete. Scored as seconds required to complete the task.
Time Frame: Baseline and Post-test at 4 weeks
Population: Elderly patients living in community nursing homes identified as fall risks with a diagnosis of probable Alzheimer's disease.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Transdermal Methylphenidate
Number analyzed (Participants) | 6
seconds
  Baseline | 34.3 (30.4)
  Post-Test | 44.2 (18.1)
Statistical Analysis 1: Comparison: Transdermal Methylphenidate; Test type: Superiority or Other; p = .55, t-test, 2 sided; Mean Difference (Final Values) = 9.9

2. Secondary Outcome: POMA -Performance Oriented Mobility Assessment - Measure of Gait and Balance.
Description: Performance Oriented Mobility Assessment (POMA), used to measure subject's ability to maintain balance. The test takes 10-15 minutes and involves asking subject to stand from a sitting position, standing with eyes closed and sitting down. POMA total score has a range of 0-36 where higher scores represent better performance. POMA total score is an additive combination of the 12 point Gait sub-score and the 16 point balance sub-score. A cut-off score of <21 is generally considered a fall risk among elderly people.
Time Frame: 4 weeks
Population: Elderly patients living in community nursing homes identified as fall risk with a diagnosis of probable Alzheimer's Disease.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Transdermal Methylphenidate
Number analyzed (Participants) | 6
Units on a scale
  Baseline | 16.7 (8.4)
  Post-Test | 17.8 (9.8)
Statistical Analysis 1: Comparison: Transdermal Methylphenidate; Test type: Superiority or Other; p = .67, t-test, 2 sided; Mean Difference (Final Values) = 1.1

ADVERSE EVENTS:
Groups:
- Single Arm Transdermal Methylphenidate: There were no adverse events reported.
Arm/Group | Single Arm Transdermal Methylphenidate
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No